CLINICAL TRIAL: NCT05940038
Title: Retrospective Study to Evaluate the Safety and Efficacy of Poly-L-l-lactic Acid [Sculptra®] in the Treatment of Skin Flaccidity in the Labia Majora and/or Pubis Region
Brief Title: Retrospective Study of the Safety and Efficacy of PLLA for Skin Flaccidity in Labia Majora and/or Pubis Region
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Galderma Brasil Ltda. (Industry)
Responsible Party: Sponsor
Other Study IDs: BR.16.003
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Phase IV, retrospective, single-center, clinical trial, chart review to evaluate the safety and efficacy of poly-L-l-lactic acid [PLLA-SCA, Sculptra®] in women who underwent at least one treatment for skin flaccidity of the labia majora and/or pubis region for safety evaluation and three treatment sessions for efficacy evaluation.

DETAILED DESCRIPTION:
This is a phase IV, retrospective, single-center, clinical trial of medical record data collection to evaluate the safety and effectiveness in subjects who have undergone at least one application of poly-L-l-lactic acid (Sculptra®) for skin flaccidity treatment in the labia majora and/or pubis region. All medical charts of subjects treated for this condition at the clinic treated from Jan1st 2022 and on will be screened for inclusion. The reason for not including a subject will be documented.

During the study, the medical records of subjects who presented skin flaccidity of the labia majora and/or pubis region will be evaluated to anamnesis and physical examination and information will be obtained on demographic data, clinical history, previous treatment(s) in the study region, number of treatment sessions with Sculptra®, as well as data on product dilution, technique used, doses injected, and adverse events related to Sculptra® and/or the injection procedure. Clinical evaluations will also be performed through the information and photographic records obtained through the evaluation of the medical records of these subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects able to read, or follow reading, understand, and sign the Informed Consent Form and the Authorization Form for Imaging Usage approved by the REC/CONEP system;
2. Subjects aged 18 years or older;
3. Having received at least 1 (one) session of Sculptra® for labia majora and/or mons pubis skin flaccidity.
4. Available clinical information and treatment data in the medical records.
5. Having medical records that present suitable photographic records prior and after the Sculptra® injections that allow a skin condition assessment of labia majora and/or mons pubis.

Exclusion Criteria:

1. Having any clinical condition or laboratory disorder, recorded at the medical record, which may compromise trial participation according to the investigator assessment.
2. Having any procedure performed on the labia majora and/or mons pubis skin within12 months prior to the first administration of PLLA (Sculptra®).
3. Participation in another clinical trial in the 30 days previous the study start.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All medical records of female subjects who received at least one (1) application of Sculptra® for the treatment of skin flaccidity of the labia majora and/or pubis, from Jan1st 2022 and on, on the private practice of the investigators will be screened for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Number of AEs | Since first application up to 12 months follow up.
Number (%) of AEs related to the study product or injection procedure | Since first application up to 12 months follow up.
Number of AEs related (%) to the study product by intensity (if available) | Since first application up to 12 months follow up.
Number (%) of subjects having at least one AE | Since first application up to 12 months follow up.
Number (%) of subjects having at least one AE related to the study product or injection procedure | Since first application up to 12 months follow up.
Number (%) of subjects who died | Since first application up to 12 months follow up.
Improvement of cutaneous flaccidity of the labia majora and/or pubis region | Since third application up to 12 months follow up since first application.
  Assessed by the percentage of total scores (n, %): hugely better, much better, or better according to Global Aesthetic Improvement Scale
Improvement of global aesthetic aspect of the labia majora and/or pubis region | Since third application up to 12 months follow up since first application.
  Assessed by the percentage of total scores (n, %): hugely better, much better, or better according to Global Aesthetic Improvement Scale

OTHER OUTCOMES:
Improvement of symptoms related to functional complaints of the labia majora and/or mons pubis region | Since third application up to 12 months follow up since first application.
  Assessed by the total percentage (n, %) of reported outcomes as hugely better, much better, or better

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Hexsel de Dermatologia, Porto Alegre, Rio Grande do Sul, Brazil